CLINICAL TRIAL: NCT07393620
Title: Predictive Value of Amplitude-Integrated Electroencephalography and Cerebral Tissue Oxygenation on Neurological Outcomes in Neonates With Mild Hypoxic-Ischemic Encephalopathy
Brief Title: Predictive Value of aEEG and Cerebral Oxygenation on Neurological Outcomes in Newborns With Mild Hypoxic-Ischemic Encephalopathy
Status: Not yet recruiting | Type: Observational
Sponsor: Uludag University (Other)
Responsible Party: Principal Investigator, Salih Çağrı Çakır, Associate professor, Uludag University
Other Study IDs: 2025/903/17-24
Record Dates: First submitted 2026-01-08; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Hypoxic-Ischemic Encephalopathy Mild
Keywords: Mild Hypoxic Ischemic Encephalopathy; Amplitude-integrated electroencephalography; Cerebral oxygenation; Near infrared spectroscopy; Neonates; aEEG; NIRS

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Newborns with mild hypoxic-ischemic encephalopathy usually do not receive cooling treatment. However, some of these newborns may develop neurological problems later in life. This observational study aims to evaluate whether early brain monitoring and measurements of brain oxygen levels are associated with neurological outcomes in newborns with mild hypoxic-ischemic encephalopathy. Newborns will be monitored during the first 72 hours after birth as part of routine clinical care. Neurological assessments will be performed during early infancy and later follow-up. The findings of this study may help improve early risk assessment and support closer monitoring of newborns who may be at increased risk for unfavorable neurological outcomes.

DETAILED DESCRIPTION:
Perinatal asphyxia resulting from impaired gas exchange may lead to hypoxemia, hypercapnia, and metabolic acidosis, causing injury to the brain and other organs in newborns. Perinatal asphyxia disrupts cerebral autoregulation, leading to primary and secondary energy deficiency, cerebral damage, and hypoxic-ischemic encephalopathy (HIE). HIE remains a significant cause of neonatal mortality and long-term neurological morbidity. HIE is clinically classified as mild, moderate, or severe based on neurological examination findings, most commonly using the Sarnat and Sarnat scoring system. Therapeutic hypothermia has been shown to reduce mortality and morbidity in term and near-term newborns with moderate to severe HIE when initiated within the first 6 hours after birth. However, therapeutic hypothermia is not routinely recommended for newborns with mild HIE due to the lack of sufficient evidence from randomized clinical trials. Although mild HIE is generally associated with a better prognosis, accumulating evidence suggests that a substantial proportion of newborns diagnosed with mild HIE may develop adverse neurodevelopmental outcomes during infancy and early childhood.

Furthermore, the severity of encephalopathy may evolve, and some newborns initially classified as having mild HIE may progress to moderate encephalopathy within the first hours after birth. Early identification of newborns with mild HIE who are at increased risk for neurological deterioration remains challenging, particularly during the critical first 6 hours of life. Continuous bedside brain monitoring techniques may provide valuable prognostic information in this early period. Amplitude-integrated electroencephalography (aEEG) allows continuous assessment of cerebral electrical activity. It helps evaluate the severity of encephalopathy, detect seizures, and predict neurological outcomes in newborns with HIE. Additionally, near-infrared spectroscopy (NIRS) allows for non-invasive monitoring of cerebral oxygenation and cerebral fractional tissue oxygen extraction (cFTOE). However, data regarding the use of NIRS in newborns with mild HIE are limited, particularly during the early postnatal period.

The primary objective of this prospective, multicenter observational cohort study is to investigate the association between early brain monitoring findings and short-term and long-term neurological outcomes in newborns with mild hypoxic-ischemic encephalopathy. Specifically, the study aims to evaluate early neurological findings and neurodevelopmental outcomes up to 24 months of age. Secondarily, this study aims to explore whether early aEEG and NIRS findings may help identify subgroups of newborns with mild HIE who are at higher risk for neurological deterioration and may benefit from closer monitoring and follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Gestational age and postnatal age:

   Gestational age ≥ 36 0/7 weeks and enrollment within the first 6 hours after birth.
2. Blood gas criteria

   Umbilical cord or postnatal (≤ 1 hour of life) blood gas showing:
   1. pH ≤ 7.00 or base deficit ≥ 16 mmol/L
   2. OR, if pH is 7.01-7.15 or base deficit is 10-15.9 mmol/L, the presence of both:

      * An acute perinatal event, and
      * Apgar score ≤ 5 at 10 minutes or ongoing resuscitation at 10 minutes of life, including the need for positive pressure ventilation.

   ( Evidence of an acute peripartum and intrapartum asphyxia event, defined by at least one of the following: Uterine rupture, placental abruption, umbilical cord prolapse, rupture, tight nuchal cord, maternal hemorrhage, trauma, or cardiopulmonary arrest, vasa previa, category III fetal heart rate tracing, including having either a sinusoidal pattern or absent baseline variability plus recurrent late decelerations, recurrent variable decelerations, or bradycardia.)
3. Clinical evidence of encephalopathy Findings consistent with Sarnat and Sarnat Stage 1 (mild) encephalopathy. Mild, moderate, or severe abnormalities may be present in at least one of the six categories (level of consciousness, spontaneous activity, posture, tone, primitive reflexes [suck and Moro], autonomic nervous system), provided that no more than two categories show moderate or severe findings.

Exclusion Criteria:

Newborns meeting any of the following criteria will be excluded from the study:

1. Normal neurological examination Newborns with a completely normal neurological examination according to Sarnat and Sarnat staging.
2. Moderate or severe encephalopathy within the first 6 hours of life

   1. Clinical findings consistent with moderate or severe encephalopathy during the first 6 hours after birth.
   2. Presence of clinical seizures.
   3. aEEG findings consistent with moderate or severe encephalopathy requiring therapeutic hypothermia.
   4. Evidence of electrographic seizure activity on aEEG monitoring.
3. Sarnat and Sarnat criteria for moderate-severe encephalopathy Findings consistent with moderate or severe encephalopathy in three or more Sarnat categories, classified as moderate or severe hypoxic-ischemic encephalopathy.
4. Contraindications to therapeutic hypothermia, including:

   * Evaluation occurring more than 6 hours after birth.
   * Gestational age < 36 weeks or birth weight < 2000 g.
   * Severe or extensive intracranial parenchymal hemorrhage.
   * Severe, life-threatening coagulopathy.
   * Intracerebral infarction.
   * Chromosomal abnormalities (e.g., trisomy 13 or 18) or major congenital anomalies involving multiple organ systems.
5. Lack of parental informed consent
6. Cyanotic congenital heart disease
7. Metabolic encephalopathy Encephalopathy due to metabolic disorders not related to hypoxic-ischemic events.
8. Other conditions associated with encephalopathy unrelated to acute hypoxia

   * Abnormal fetal growth.
   * Maternal infections.
   * Fetomaternal hemorrhage.
   * Severe neonatal sepsis.
   * Chronic placental lesions.

Ages: 0 Hours to 6 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study population consists of newborns with a gestational age of ≥ 36 0/7 weeks who are diagnosed with mild hypoxic-ischemic encephalopathy within the first 6 hours after birth. Eligible participants include newborns with evidence of an acute peripartum or intrapartum asphyxial event who meet blood gas and clinical criteria for hypoxic-ischemic injury but do not fulfill criteria for moderate or severe encephalopathy or for therapeutic hypothermia at enrollment. Newborns will be prospectively followed from birth up to 24 months of age to assess both short-term and long-term neurological outcomes.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2026-02-10 (Estimated); Primary Completion 2027-02-10 (Estimated); Study Completion 2029-02-10 (Estimated)

PRIMARY OUTCOMES:
Neurological Outcomes in Neonates with Mild Hypoxic-ischemic Encephalopathy | at 18 and 24 months of age
  The primary outcome measure is the report of neurological outcome in children diagnosed with mild hypoxic-ischemic encephalopathy. Neurological outcome will be measured using the Bayley Scales of Infant and Toddler Development (Bayley-III) at 18-24 months of age; a standard score below 85 in at least one of the cognitive, motor, or language domains will be defined as a neurologic disorder.

SECONDARY OUTCOMES:
Correlation Between Early aEEG Background Patterns and Neurological Outcomes in Newborns With Mild Hypoxic-Ischemic Encephalopathy | aEEG: within the first 72 hours of life. Neurological outcomes: at 18 and 24 months of age, birth to 24 months of age.
  This outcome measure evaluates the correlation between:
  1. Continuous amplitude-integrated electroencephalography (aEEG) monitoring will be used within the first 72 hours of life to measure the amplitude (µV) of cerebral electrical activity and to determine background patterns and sleep-wake cycling; and
  2. Neurological outcomes, measured by the Bayley Scales of Infant and Toddler Development (Bayley-III) in the cognitive, motor, and language domains at 18 and 24 months of age.
Correlation Between Early Cerebral NIRS Values and Neurological Outcomes in Newborns With Mild Hypoxic-Ischemic Encephalopathy | Cerebral NIRS: within the first 72 hours of life. Neurological outcomes: at 18 and 24 months of age, birth to 24 months of age.
  This outcome measure evaluates the correlation between:
  1. Early cerebral NIRS values within the first 72 hours of life. Cerebral oxygenation (%) values at NIRS measurements in infants, first 6 h of life, first 24 h of life, between 24-48 h, 48-72 h.
  2. Neurological outcomes, measured by the Bayley Scales of Infant and Toddler Development (Bayley-III) in the cognitive, motor, and language domains at 18 and 24 months of age.

CONTACTS AND LOCATIONS:
Locations (3):
- Turkey (Türkiye) (3):
  - Bursa City Hospital, Bursa
  - Division of Neonatology, Department of Pediatrics, Bursa Uludağ University Faculty of Medicine, Bursa
  - Division of Neonatology, Department of Pediatrics, University of Health Sciences Bursa Yuksek İhtisas Training and Research Hospital, Bursa

IPD SHARING:
Plan to Share IPD: No
I am not authorized to share patient data.

REFERENCES:
- [Background] Shalak LF, Laptook AR, Velaphi SC, Perlman JM. Amplitude-integrated electroencephalography coupled with an early neurologic examination enhances prediction of term infants at risk for persistent encephalopathy. Pediatrics. 2003 Feb;111(2):351-7. doi: 10.1542/peds.111.2.351. PMID 12563063
- [Background] Chalak L. New Horizons in Mild Hypoxic-ischemic Encephalopathy: A Standardized Algorithm to Move past Conundrum of Care. Clin Perinatol. 2022 Mar;49(1):279-294. doi: 10.1016/j.clp.2021.11.016. Epub 2022 Jan 21. PMID 35210007
- [Background] Kariholu U, Montaldo P, Markati T, Lally PJ, Pryce R, Teiserskas J, Liow N, Oliveira V, Soe A, Shankaran S, Thayyil S. Therapeutic hypothermia for mild neonatal encephalopathy: a systematic review and meta-analysis. Arch Dis Child Fetal Neonatal Ed. 2020 Mar;105(2):225-228. doi: 10.1136/archdischild-2018-315711. Epub 2018 Dec 19. PMID 30567775
- [Background] Chalak LF, Nguyen KA, Prempunpong C, Heyne R, Thayyil S, Shankaran S, Laptook AR, Rollins N, Pappas A, Koclas L, Shah B, Montaldo P, Techasaensiri B, Sanchez PJ, Sant'Anna G. Prospective research in infants with mild encephalopathy identified in the first six hours of life: neurodevelopmental outcomes at 18-22 months. Pediatr Res. 2018 Dec;84(6):861-868. doi: 10.1038/s41390-018-0174-x. Epub 2018 Sep 13. PMID 30250303
- [Background] Prempunpong C, Chalak LF, Garfinkle J, Shah B, Kalra V, Rollins N, Boyle R, Nguyen KA, Mir I, Pappas A, Montaldo P, Thayyil S, Sanchez PJ, Shankaran S, Laptook AR, Sant'Anna G. Prospective research on infants with mild encephalopathy: the PRIME study. J Perinatol. 2018 Jan;38(1):80-85. doi: 10.1038/jp.2017.164. Epub 2017 Nov 2. PMID 29095433
- [Background] Conway JM, Walsh BH, Boylan GB, Murray DM. Mild hypoxic ischaemic encephalopathy and long term neurodevelopmental outcome - A systematic review. Early Hum Dev. 2018 May;120:80-87. doi: 10.1016/j.earlhumdev.2018.02.007. Epub 2018 Feb 26. PMID 29496329
- [Background] Murray DM, O'Connor CM, Ryan CA, Korotchikova I, Boylan GB. Early EEG Grade and Outcome at 5 Years After Mild Neonatal Hypoxic Ischemic Encephalopathy. Pediatrics. 2016 Oct;138(4):e20160659. doi: 10.1542/peds.2016-0659. Epub 2016 Sep 20. PMID 27650049